CLINICAL TRIAL: NCT03345810
Title: Durvalumab (MEDI4736) in Frail and Elder Patients With Metastatic NSCLC (DURATION)
Acronym: DURATION
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AIO-Studien-gGmbH (Other)
Collaborators: AstraZeneca (Industry); Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIO-YMO/TRK-0416; 2016-003963-20 (EudraCT Number); ESR-15-11003 (Other Grant/Funding Number: AstraZeneca GmbH); AX-CL-NSCLC-AIO-008260 (Other Grant/Funding Number: Celgene)
Record Dates: First submitted 2017-11-14; First posted 2017-11-17 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Metastatic Lung Cancer; Non Small Cell Lung Cancer; Lung Adenocarcinoma Metastatic; Large Cell Lung Carcinoma Metastatic
Keywords: NSCLC; Non small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — durvalumab; Vinorelbine; Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Arm A (Active Comparator): Frail or elderly patients with metastatic NSCLC; CARG- Score ≤ 3 Carboplatin (AUC 5.0; D1) + nab-Paclitaxel (100mg/m2 D1,D8) Q3W
  Interventions: Drug: nab-Paclitaxel; Drug: Carboplatin
- Experimental Arm B (Experimental): Frail or elderly patients with metastatic NSCLC; CARG- Score ≤ 3
  Induction:Carboplatin (AUC 5.0; D1) + nab-Paclitaxel (100mg/m2) D1,D8; Q3W [2 cyc] followed by durvalumab (1125 mg; Q3W) [ 2 cyc] Maintenance:durvalumab (1500 mg) Q4W
  Interventions: Drug: Durvalumab; Drug: nab-Paclitaxel; Drug: Carboplatin
- Experimental Arm C (Experimental): Frail or elderly patients with metastatic NSCLC; CARG- Score > 3
  Induction: Vinorelbine (30 mg/m2; D1+D8) Q3W [ 2 cyc] or Gemcitabine (1000 mg/m2; D1+D8) Q3W [ 2 cyc] followed by durvalumab (1125 mg) Q3W [2 cyc] Maintenance:durvalumab (1500 mg; Q4W)
  Interventions: Drug: Durvalumab; Drug: Vinorelbine; Drug: Gemcitabine
- Control Arm D (Active Comparator): Frail or elderly patients with metastatic NSCLC; CARG- Score > 3
  Vinorelbine (30 mg/m2; D1+D8) Q3W or Gemcitabine (1000 mg/m2; D1+D8) Q3W
  Interventions: Drug: Vinorelbine; Drug: Gemcitabine

INTERVENTIONS:
Drug: Durvalumab — Induction: (1125 mg) cycle Q3W Maintenance: (1500 mg) cycle Q4W
  Other Names: MEDI4736
  Arms: Experimental Arm B; Experimental Arm C
Drug: Vinorelbine — (30 mg/m2 D1 + D8 as infusion) cycle Q3W
  Arms: Control Arm D; Experimental Arm C
Drug: Gemcitabine — (1000 mg/m2 D1 + D8 as infusion) cycle Q3W
  Arms: Control Arm D; Experimental Arm C
Drug: nab-Paclitaxel — (100 mg/m2 intravenous infusion over 30 minutes on D1, D8) cycle Q3W
  Other Names: Abraxane
  Arms: Control Arm A; Experimental Arm B
Drug: Carboplatin — (AUC = 5 mg•min/mL on Day 1) cycle Q3W
  Arms: Control Arm A; Experimental Arm B

SUMMARY:
AIO-YMO/TRK-0416 (DURATION) is a open-label, treatment stratified and randomized phase II study of Durvalumab, frail or elderly patients with metastatic non-squamous NSCLC with no targetable molecular alterations (EGFRwt; ALKtransl-) and not amenable to cisplatinum-based standard-combination chemotherapy but eligible for at-least mono-chemotherapy with gemcitabine or vinorelbine.

DETAILED DESCRIPTION:
The primary objective is to assess the safety and tolerability of sequential therapy consisting of standard of care mono- or combination chemotherapy followed by durvalumab in comparison to standard of care mono- or combination chemotherapy in frail/elderly patients.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and any locally-required authorization (EU Data Privacy Directive in the EU) obtained from the subject prior to performing any protocol-related procedures, including screening evaluations
2. Age ≥ 70 years at time of study entry and/or Charlson-Comorbidity-Index (CCI) >1 and/or Performance status ECOG >1
3. Histologically confirmed diagnosis of metastatic NSCLC and no targetable molecular alterations (EGFRwt; ALKtransl-) and not amenable to cisplatinum-based standard-combination chemotherapy.
4. Patients with measurable disease (at least one uni-dimensionally measurable target lesion not previously irradiated, by CT-scan or MRI) according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1) are eligible.
5. A formalin fixed, paraffin-embedded (FFPE) tumor tissue block (fresh or archival less than 3 years old or recent) or a minimum of 10 unstained slides of tumor sample (slices must be less than 90 days old and collected on SuperFrost slides provided by the sponsor) must be available for biomarker (PD-L1) evaluation. Biopsy should be excisional, incisional or core needle. Fine needle aspiration is inappropriate.
6. No prior chemotherapy or any other systemic therapy for metastatic NSCLC. Patients who have received prior platinum-containing adjuvant, neoadjuvant, or definitive chemoradiation for locally advanced disease are eligible, provided that progression has occurred >6 months from last therapy.
7. Prior radiotherapy and surgery are allowed if completed 4 weeks (for minor surgery and palliative radiotherapy for bone pain: 2 weeks) prior to start of treatment and patient recovered from toxic effects or associated adverse events.
8. Adequate blood count, liver-enzymes, and renal function:

   * Haemoglobin ≥ 9.0 g/dL
   * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L (> 1500 per mm3)
   * Platelet count ≥ 100 x 109/L (>100,000 per mm3)
   * Serum bilirubin ≤ 1.5 x ULN. This will not apply to subjects with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.
   * AST (SGOT)/ALT (SGPT) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be ≤ 5x ULN
   * Serum creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance
9. Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits, examinations including follow up and appropriate contraception

Exclusion Criteria:

1. Mixed small-cell lung cancer and NSCLC histology
2. Mean QT interval corrected for heart rate (QTc) ≥470 ms calculated from 3 electrocardiograms (ECGs) using Fredericia's correction
3. History of another primary malignancy except local prostate cancer without need for systemic treatment (e.g. active surveillance, operation without need for adjuvant treatment) and malignancies treated with curative intent and with no known active disease >2 years befor the first dose of study drug and of low potential risk for recurrence, e.g. adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease, adequately treated carcinoma in situ without evidence of disease (e.g. cervical cancer in situ)
4. Pre-existing peripheral neuropathy of Grade ≥ 2
5. Brain metastasis or spinal cord compression unless asymptomatic or treated and stable off steroids and anti-convulsants for at least 1 month prior to study treatement.
6. Active or prior documented autoimmune disease within the past 2 years. NOTE: Subjects with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded.
7. Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis)
8. History of primary immunodeficiency
9. History of allogeneic organ transplant
10. History of hypersensitivity to durvalumab or any excipient
11. History of hypersensitivity to any of the comparator agents
12. Medication that is known to interfere with any of the agents applied in the trial.
13. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses including any subject known to have evidence of acute or chronic hepatitis B, hepatitis C or human immunodeficiency virus (HIV), or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent
14. Clinical diagnosis of active tuberculosis
15. Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving durvalumab
16. Male patients of reproductive potential who are not employing an effective method of birth control (failure rate of less than 1% per year)
17. Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results
18. Participation in another clinical study with an investigational product during the last 30 days before inclusion
19. Any previous treatment with a PD-1 or PD-L1 inhibitor, including durvalumab
20. Current or prior use of immunosuppressive medication within 28 days before the first dose of durvalumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid
21. Receipt of the last dose of anti-cancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies, other investigational agent) ≤ 21 days prior to the first dose of study drug or ≤4 half-lifes of the agent administered, which ever comes first.
22. Previous enrollment or randomization in the present study.
23. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff of sponsor and study site)
24. Patient who might be dependent on the sponsor, site or the investigator
25. Patient who has been incarcerated or involuntarily institutionalized by court order or by the authorities § 40 Abs. 1 S. 3 Nr. 4 AMG.
26. Patients who are unable to consent because they do not understand the nature, significance and implications of the clinical trial and therefore cannot form a rational intention in the light of the facts [§ 40 Abs. 1 S. 3 Nr. 3a AMG].

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-12-14 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Rate of treatment related Grade III/IV adverse events (CTCAE V4.03) | through study completion, an average of 24 months
  Comparison of the outcome of sequential therapy consisting of standard of care mono- or combination chemotherapy followed by durvalumab versus standard of care mono- or combination chemotherapy in frail/elderly patients

SECONDARY OUTCOMES:
PFS | approx. 24 months
  Progression Free Survival
ORR using assessment according to RECIST 1.1 | approx. 24 months
  Response Evaluation Criteria In Solid Tumors (RECIST)
OS | approx. 60 months
  Overall Survival
Adverse Events /Serious Adverse Events | approx. 48 months
  Adverse Events: Type, incidence, and severity according to NCI CTCAE version 4.03
Health related Quality of Life (HR-QoL) | approx. 60 months
  as determined with FACT-L (Functional Assessment of Cancer Therapy - Lung)
Geriatric assessment | approx. 60 months
  G8-questionnaire
Geriatric assessment | approx. 60 months
  Timed up & go (test of basic functional mobility)
Geriatric assessment | approx. 60 months
  6MWT (6 minutes walk test)

CONTACTS AND LOCATIONS:
Overall Officials: Jonas Kuon, Dr, Principal Investigator — Department of Thoracic Oncology, Thoraxklinik at Heidelberg University Hospital, Heidelberg, Germany
Locations (30):
- Germany (30):
  - Gesundheitszentrum St. Marien GmbH, Amberg
  - Ev. Lungenklinik Berlin, Berlin
  - Kliniken der Stadt Köln gGmbH, Cologne
  - Klinikum Darmstadt, Darmstadt
  - Universitätsklinikum Carl-Gustav-Carus, Dresden
  - Klinikum Esslingen, Esslingen am Neckar
  - Universitätsklinikum Frankfurt, Frankfurt am Main
  - Klinik Schillerhöhe, Gerlingen
  - Universitätsmedizin Greifswald, Greifswald
  - Onkodoc GmbH, Gütersloh
  - Krankenhaus Martha-Maria Halle Dölau, Halle
  - Department of Thoracic Oncology, Thoraxklinik at Heidelberg University Hospital, Heidelberg
  - Lungenklinik Hemer, Hemer
  - "Vincentius-Diakonissen-Kliniken gAG, Karlsruhe
  - Ortenau-Klinikum Lahr, Lahr
  - Ev. Diakonissenkrankenhaus Leipzig, Leipzig
  - Klinik Löwenstein gGmbH, Löwenstein
  - Klinikum Ludwigsburg, Ludwigsburg
  - DRK-Kliniken Berlin Mitte, Mitte
  - Klinikum der Universität München, München
  - Pius Hospital Oldenburg, Oldenburg
  - Krankenhaus Barmherzige Brüder, Regensburg
  - "Klinikum Rheine, Rheine
  - Marienhospital, Stuttgart
  - Krankenhaus der Barmherzigen Brüder, Trier
  - Universitätsklinikum Ulm, Ulm
  - Schwarzwald-Baar Klinikum, Villingen-Schwenningen
  - SHG-Kliniken-Völklingen, Völklingen
  - Hämatologisch-Onkologische Praxis Würselen, Würselen
  - Klinikum Würzburg Mitte gGmbH, Würzburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kuon J, Hommertgen A, Krisam J, Lasitschka F, Stenzinger A, Blasi M, Bozorgmehr F, Maenz M, Kieser M, Schneider M, Thomas M. Durvalumab in frail and elderly patients with stage four non-small cell lung cancer: Study protocol of the randomized phase II DURATION trial. Trials. 2020 Apr 22;21(1):352. doi: 10.1186/s13063-020-04280-8. PMID 32321565
- See also: AIO - Working Group for Medical Oncology from the German Cancer Society — http://www.aio-portal.de
- See also: AIO-Studien-gGmbH — http://www.aio-studien-ggmbh.de